CLINICAL TRIAL: NCT04763603
Title: Assessment of Plaque Vulnerability Using a Novel Technique: Multi-spectral PhotoAcoustic Imaging.
Acronym: (CVENT-PAI)
Status: Terminated | Type: Observational
Why Stopped: SARS-CoV-2 coronavirus outbreak and end of funding
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D18-P007
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Neurology
Keywords: carotid stenosis; Photoacoustic imaging; Laser diode
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — atherosclerotic plaque
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identification of intraplaque haemorrhage using MRI is technically demanding and sometimes uncomfortable. Photoacoustic imaging is a new non-invasive technique combining multi-wavelength infrared laser light and ultrasound imaging, able to discriminate blood and other components in the tissues. The measurement by the multi-spectral photoacoustic imaging is likely to be more acceptable and therefore could replace MRI.

DETAILED DESCRIPTION:
A total of 60 patients with stenosis grade of > 70% and considered for endarterectomy will be recruited for additional imaging. Pre-operative PA/US and 3D MR imaging will be conducted. Two patient groups are designed to allow performance assessment with respect to anatomy, i.e., penetration depth; One with favourable anatomy (i.e. superficial carotids, proximal plaques and low bifurcation), the other with no anatomical considerations. For in-vivo verification of the morphology and mechanical properties obtained with PA/US imaging, the pre-operative data will be compared to the MR data (imaging-imaging verification). Since the patient is operated on, endarterectomy specimens are available for histo-pathological examination and in-vitro testing for verification purposes: the excised tissue will be (snap freeze with liquid Nitrogen) transported to TUE in Eindhoven for in-vitro validation (imaging-histology verification). Paris patients will undergo surgery and tissues will be transferred to Eindhoven for in vitro mechanical testing. Because of the transfer (-80 °C), the rate of success for in vitro testing is expected to be smaller, around 40% (i.e. 12 subjects). Nevertheless, the power of the global analysis will be increased.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one carotid plaque with a degree of stenosis 70% (NASCET), indication to surgery (endarterectomy),
* Patients with favourable anatomy criteria :

x Cranio-caudal length of normal or long neck x Cervical adiposity weak or absent x Carotid bifurcation in usual situation (at the level of the mandibular angle or lower) x Normal genicity of subcutaneous tissues x Calcification of arterial moderate or absent

* Patients affiliated to the social health security system.

Exclusion Criteria:

* Refusal to participate,
* any concomitant chronic condition hampering the realization of ultrasound scanner or MRI (allergy to gel, intolerance or contraindication to gadolinium).
* Unstable patients with plaque claudication inducing procedure acceleration.
* Patients with unfavourable anatomy criteria :

x Cranio-caudal length of the neck very short x Significant cervical adiposity x Carotid bifurcation higher than the mandibular angle x High echogenic subcutaneous tissue x Calcification marked arterialH2020-ICT-29-2016 no. 731771 Ethics requirements x Patients with fat necks, Presence of extensive calcifications at the site of the stenosis.

* Patients unable to consent.
* Pregnant woman or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project involves patients with atherosclerotic plaques (either symptomatic or not).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of the device | 18 month
  The primary outcome is to evaluate the ability of the experimental device to visualize hemorrhage within the plaque. The primary endpoint will therefore be concordance with histology and plaque analysis (ex-vivo reference method) and MRI (invivo reference method).

SECONDARY OUTCOMES:
Evaluation of anatomical concordance | 18 month
  The secondary objective of the study is to evaluate the concordance according to the anatomical characteristics of the patient. However, only patients without unfavorable anatomy will be included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Anne Hospital, Paris, Île-de-France Region, France

REFERENCES:
- See also: Cvent projet website — https://cvent-2020.eu/project.html